CLINICAL TRIAL: NCT06930638
Title: MitoQ and Ischemic Conditioning To Assess Vascular Health Outcomes (MITO Study)
Brief Title: MitoQ and Ischemic Conditioning To Assess Vascular Health Outcomes
Acronym: MITO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: PRO00054821
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: Ischemic Conditioning; Blood Flow; Microvascular Health; Flow-Mediated Dilation; Antioxidant; Reactive Oxygen Species; Supplement
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Ischemic Conditioning - High (Experimental): During each testing session, the investigators will be measuring how one treatment of ischemic conditioning affects blood flow and muscle function. One day participants will receive a high cuff inflation pressure on the leg, called ischemic conditioning - high (225 mmHg).
  Interventions: Device: Ischemic Conditioning
- Ischemic Conditioning - Low (Experimental): During each testing session, the investigators will be measuring how one treatment of ischemic conditioning affects blood flow and muscle function. One day participants will receive a low cuff inflation pressure on the leg, called ischemic conditioning - low (25 mmHg).
  Interventions: Device: Ischemic Conditioning
- Antioxidant Supplement (Experimental): During each testing session, the investigators will be measuring how one treatment of an over-the-counter antioxidant supplement affects blood flow and muscle function. One day participants will orally ingest an over-the-counter antioxidant supplement called MitoQ.
  Interventions: Dietary Supplement: Antioxidant Supplement

INTERVENTIONS:
Device: Ischemic Conditioning — The cuff will be placed around the proximal, non-affected thigh and inflated for 5 minutes in a supine or semi-reclined position, then released for a 5-minute recovery period. Five cycles of inflation and recovery will be performed (45 minutes total).These inflations will be done using a cuff similar to what is used for taking blood pressure.
  Arms: Ischemic Conditioning - High; Ischemic Conditioning - Low
Dietary Supplement: Antioxidant Supplement — MitoQ is an over the counter supplement that increases delivery to the mitochondria. Similar to studies performed in middle age/older adults and individuals with peripheral arterial disease, we will administer 1 single oral dose of 80mg of MitoQ or a placebo pill. As MitoQ reaches peak concentrations at ~40 to 60 minutes after ingestion, we will wait 45 minutes (time matched to Ischemic conditioning).
  Arms: Antioxidant Supplement

SUMMARY:
Stroke survivors have compromised vascular function which may contribute to secondary stroke risk, cardiovascular disease, and may limit their exercise tolerance. Preliminary data shows a single bout of ischemic conditioning or oral ingestion of an over-the-counter antioxidant supplement called MitoQ may improve vascular function and muscle activity in individuals post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years of age
* Cortical or sub-cortical stroke ≥ 6 months ago with residual hemiparesis
* Able to give informed consent and follow 2-step command.
* English Speaking

Exclusion Criteria:

* Unable to stand from chair without physical assistance from another person (able to use assistive device).
* History of blood clots in the extremities or any condition in which compression of the thigh or transient ischemia is contraindicated (i.e., wounds in the leg).
* Chronic lasting symptoms (> 6 months) of severe COVID-19 (i.e., hospitalization)
* History of head trauma or concussion within the past 6 months
* Comorbid neurological disorder
* Peripheral vascular disease
* Myocardial infarction or arrhythmia in the previous year
* Resting SBP ≥180 mmHg or DBP ≥ 100 mmHg
* Pregnant or breastfeeding.
* Other significant medical condition likely to influence study or jeopardize safety as assessed by the Primary Investigator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Brachial Artery Flow-Mediated Dilation | Change from BL to Post Intervention (5 hours)
  We will measure brachial artery vascular health in the non-paretic arm. Baseline brachial artery diameter and blood flow velocity through the artery will be measured before and after a pneumatic forearm cuff is inflated to 225 mmHg for five minutes.
Microvascular Vasodilation | Change from BL to Post Intervention (5 hours)
  Laser Doppler Flowmetry (LDF) with Dermal Microdialysis (DM) will measure blood flow flux during microinfusions of study drugs (limited to an area on the skin approximately the size of a nickel) to examine endothelial dependent vasodilation (Acetylcholine, ACh) and nitric-oxide mediated vasodilation (ACH +/- LNAME, and endothelial nitric oxide synthase inhibitor).

SECONDARY OUTCOMES:
Muscle Tissue Oxygenation | Change from BL to Post Intervention (5 hours)
  We will also place a near-infrared spectroscopy (NIRS) pad on the thenar eminence of the non-paretic hand to non-invasively measure tissue oxygenation via infrared light following the pneumatic forearm cuff inflation/deflation.
Blood Draw | Change from BL to Post Intervention (5 hours)
  We will collect blood before and after the intervention via an in-dwelling intravenous catheter. The blood draw analysis may include but will not be limited to examining complete blood counts, glucose levels, cholesterol, and plasma redox and bioenergetic analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Durand, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No